CLINICAL TRIAL: NCT01528592
Title: A Pilot Study of the Drug Effects on Brain Connectivity of Parkinson's Disease
Brief Title: PharmacoMRI of Parkinson Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Darren Gitelman, Medical Doctor, Associate Professor of Neurology and Physiology, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Ruby-60029592
Record Dates: First submitted 2012-01-31; First posted 2012-02-08 (Estimated); Results first posted 2013-12-24 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-04

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — carbidopa, levodopa drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- On / Off medication (Experimental): Subjects undergo MRI scanning in the medication off state and 1 hour after receiving medications.
  Interventions: Drug: Carbidopa-Levodopa

INTERVENTIONS:
Drug: Carbidopa-Levodopa — Equivalent amount of carbidopa-levodopa will be provide to you

SUMMARY:
Based on studies showing better responsiveness of motor versus cognitive symptoms to Parkinson's Disease medication, also known as dopaminergic treatments, the investigators hypothesize that comparison of resting state networks in the on versus off medication state in Parkinson's Disease patients will show greater effects on brain networks associated with motor control.

DETAILED DESCRIPTION:
Subject participation includes two 25-30 minute MRI scans. The subject will arrive in the "off" state (PD medications withheld for approximately 12 hours prior to the scan). Following the initial scan, the subject will receive 125% of his or her usual daily morning dose of PD medications which is calculated as levodopa dose equivalents (LDE) and is given as carbidopa-levodopa. The subject will then wait for an hour allowing for the medication to begin working. During this time the subject will complete cognitive assessments, questionnaires regarding the history and current state of PD, and motor assessments. The subject will then undergo a second MRI scan of approximately 25-30 minutes. The subject after completing the second MRI scan is free to leave. The entire study is approximately 2 and 1/2 hours long.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's Disease (PD)
* Older than 30 years of age at the time of diagnosis
* Hoehn and Yahr stage greater than or equal to 2.5
* PD duration greater than 3 years
* Stable regimen of PD medications for at least 2 weeks prior to imaging
* PD medications include carbidopa-levodopa

Exclusion Criteria:

* Patients with a diagnosis of other neurodegenerative conditions
* Patients unwilling or unable to give informed consent
* Contraindications (cardiac pacemaker, etc.) or inability (e.g., claustrophobia) to undergo MRI scan

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-06; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darren R Gitelman, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: 12/1/2011 - 4/30/2012 Location: Medical clinic in Chicago
Period: Overall Study
Arm/Group | On / Off Medication
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients with Parkinson's disease on dopaminergic therapy.
Arm/Group | On / Off Medication
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.22 (8.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Correlation Coefficient Between UPDRS III Score and Independent Components Analysis Network Strength in Left Parietal Cortex.
Description: Correlation coefficient between UPDRS III score and independent components analysis network strength in left parietal cortex. UPDRS III is the Unified Parkinson's Disease Rating Scale composite motor score.
Time Frame: 1 hour
Measure: Number; unit: unitless
Arm/Group | On / Off Medication
Number analyzed (Participants) | 15
unitless | 0.5869

ADVERSE EVENTS:
Arm/Group | On / Off Medication
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No